CLINICAL TRIAL: NCT04902170
Title: The Surgical Outcomes of Long-shaft Vitrectomy Probe for Vitreoretinal Diseases in Highly Myopic Eyes
Brief Title: Long-shaft Vitrectomy Probe in Highly Myopic Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202008057DIFD
Record Dates: First submitted 2021-02-21; First posted 2021-05-26 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2021-11

CONDITIONS: Retinal Diseases; High Myopia
Keywords: High myopia; Pars plana vitrectomy; Vitreoretinal disease
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Highly myopic patients with vitreoretinal disease requiring pars plana vitrectomy. The 30mm (shaft length) vitrectomy probe (25 gauge) would be used in the surgery.
  Interventions: Procedure: 25 gauge pars plana vitrectomy
- control group (Active Comparator): Highly myopic patients with vitreoretinal disease requiring pars plana vitrectomy. The 27mm (shaft length) vitrectomy probe (25 gauge) would be used in the surgery.
  Interventions: Procedure: 25 gauge pars plana vitrectomy

INTERVENTIONS:
Procedure: 25 gauge pars plana vitrectomy — 25 gauge pars plana vitrectomy

SUMMARY:
This study aimed to compare the safety and efficacy of vitrectomy probe with different shaft lengths in vitreoretinal surgery of highly myopic patients. In this randomized controlled study, highly myopic patients who had axial length more than 26 mm and needed vitreoretinal surgery will be enrolled. The enrolled patients will be randomized into "30 mm shaft length group"(trial group) and "27mm shaft length group"(controlled group). We will compare the rate of wound leakage, hypotony, subconjunctival hemorrhage, probe bending, trocar removal, and endophthalmitis between the two groups. We would like to evaluate the efficacy and safety of the 30 mm shaft length vitrectomy probe.

ELIGIBILITY:
Inclusion Criteria:

* Highly myopic patients (axial length > 26mm) with vitreoretinal diseases or maculopathy requiring pars plana vitrectomy

Exclusion Criteria:

* Previous history of pars plana vitrectomy
* Surgical plan combining encircling buckle
* Silicone oil or perfluorocarbon liquid use intraoperatively
* Previous history of pterygium surgery, trabeculectomy, glaucoma surgery
* Previous history of corneal, conjunctival, or scleral laceration
* History of connective tissue disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
trocar removal rate | intra-operative
  trocar removal would be performed if the length of vitrectomy probe was not adequate
operation time | intra-operative
  record the operation time and time of core vitrectomy

SECONDARY OUTCOMES:
instrument bending | intraoperative
  record the occurrence of instrument bending

OTHER OUTCOMES:
Complications | Until post-op 6 month
  the presence of vitreous hemorrhage, retinal hemorrhage, retinal detachment, choroidal hemorrhage, endophthalmitis
wound status evaluation by slit lamp biomicroscopy | until post-op 1 month
  the presence of subconjunctival hemorrhage, chemosis, subconjunctival air, wound suture
anatomical success evaluation by optical coherence tomography and indirect ophthalmolscopy | post-op 3 month
  whether the disease was successfully treated
anatomical success evaluation by optical coherence tomography and indirect ophthalmolscopy | post-op 6 month
  whether the disease was successfully treated

CONTACTS AND LOCATIONS:
Overall Officials: Tzyy-Chang Ho, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan